CLINICAL TRIAL: NCT04067830
Title: Preoperative Respiratory Muscle Training to Prevent Postoperative Pulmonary Complications in Patients Undergoing Resection for Lung Cancer
Brief Title: Respiratory Muscle Training Before Surgery in Preventing Lung Complications in Patients With Stage I-IIIB Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I 72818; NCI-2019-03537 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 72818 (Other: Roswell Park Cancer Institute); R01CA222382 (NIH)
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Laparoscopy; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm I (usual care) (Active Comparator): Patients receive usual care consisting of physical therapy once weekly, receiving pre-surgical information, instruction on the use of a spirometer device, and wearing a Fitbit to track activity. Patients then undergo video-assisted thoracic surgery or laparoscopic surgery. Patients continue to track activity using the Fitbit for 3 months post-surgery.
  Interventions: Other: Best Practice; Procedure: Laparoscopic Surgery; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Video-Assisted Thoracic Surgery
- Arm II (RMT + usual care) (Experimental): Patients use a power lung device to complete 3 sets of 15 RMT exercises over 30 minutes 6 days per week over 2-4 weeks for a minimum of 12 sessions prior to surgery. Patients also receive usual care consisting of attending physical therapy once weekly, receiving pre-surgical information, instruction on the use of a spirometer device, and wearing a Fitbit to track activity. Patients then undergo video-assisted thoracic surgery or laparoscopic surgery. Patients continue to track activity using the Fitbit for 3 months post-surgery.
  Interventions: Other: Best Practice; Procedure: Laparoscopic Surgery; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Device: Respiratory Muscle Training Device; Procedure: Video-Assisted Thoracic Surgery

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
Procedure: Laparoscopic Surgery — Undergo laparoscopic surgery
  Other Names: laparoscopic-assisted resection; laparoscopy-assisted surgery
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Device: Respiratory Muscle Training Device — Use power lung device to complete RMT
  Arms: Arm II (RMT + usual care)
Procedure: Video-Assisted Thoracic Surgery — Undergo video-assisted thoracic surgery
  Other Names: VATS

SUMMARY:
This phase II trial studies how well respiratory muscle training before surgery works in preventing lung complications after surgery in patients with stage I-IIIB lung cancer. Patients with lung cancer who choose to undergo surgical resection often have complications after surgery such as pneumonia, unplanned intubations, difficulty breathing and reduced physical functioning, and increased medical costs and a reduced quality of life. Improving pre-surgical pulmonary health through respiratory muscle training may improve respiratory muscle strength, response to surgery, and quality of life after surgery in patients with lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the impact of a short-duration respiratory muscle training (RMT) program on respiratory muscle strength in patients undergoing resection for lung cancer.

SECONDARY OBJECTIVES:

I. Compare the extent of diaphragm atrophy and catabolic/anabolic pathway activation between RMT responders and non-responders evaluated for gene expression and candidate and candidate causative protein levels.

II. Determine the effect of the short-duration RMT program on health related quality-of-life measures.

III. Assess the impact of the short-duration RMT program on postoperative outcomes.

EXPLORATORY OBJECTIVES:

I. Determine the financial sustainability of a transitional home-based prehabilitation program targeting respiratory muscle weakness prior to lung resection.

II. Analysis of molecular markers to correlate with patient outcome and potentially differentiate responders from non-responders.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (USUAL CARE): Patients receive usual care consisting of physical therapy once weekly, receiving pre-surgical information, instruction on the use of a spirometer device, and wearing a Fitbit to track activity. Patients then undergo video-assisted thoracic surgery or laparoscopic surgery. Patients continue to track activity using the Fitbit for 3 months post-surgery.

ARM II (RMT + USUAL CARE): Patients use a power lung device to complete 3 sets of 15 RMT exercises over 30 minutes 6 days per week over 2-4 weeks for a minimum of 12 sessions prior to surgery. Patients also receive usual care consisting of physical therapy once weekly, receiving pre-surgical information, instruction on the use of a spirometer device, and wearing a Fitbit to track activity. Patients then undergo video-assisted thoracic surgery or laparoscopic surgery. Patients continue to track activity using the Fitbit for 3 months post-surgery.

After completion of study, patients are followed up at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented stage I-IIIb lung cancer or is undergoing surgery for diagnosis
* Participant is able to speak, read, and comprehend English
* Participant must be undergoing or is anticipated to either video-assisted thoracic surgery (VATS or robotic surgery) or laparoscopic surgery for curative intent lung resection
* Patients with or without neoadjuvant chemoradiotherapy (CRT) prior to surgery will be included
* Ability to follow written and verbal instructions
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Documented ischemic heart disease; congestive heart failure or; significant cardiac arrhythmias that would exclude them from having surgery
* Overall medical frailty (clinician discretion) or ECOG > 2
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2027-03-22 (Estimated); Study Completion 2027-03-22 (Estimated)

PRIMARY OUTCOMES:
Change in inspiratory and expiratory muscle strength | Baseline up to 12 months
  Will be treated as a continuous variable and will be summarized by treatment group and time-point using the mean, median, standard deviation, and the appropriate percentiles. The effectiveness of the respiratory muscle training (RMT) program on each respiratory outcome will be assessed by comparing the preoperative change between groups using an analysis of covariance (ANCOVA) model, with an adjustment for the pretreatment levels. For each outcome, the preoperative change (T1-T0) will be modeled as a function of treatment group (RMT versus usual care) and pre-treatment levels. A one-sided Wald type-test about coefficient for treatment group will evaluate whether the RMT program had a beneficial impact on the given respiratory outcome. All model assumptions will be verified graphically using quantile-quantile and residual plots. Transformations will be applied as appropriate.
Change in pulmonary function and respiratory muscle endurance | Baseline up to 12 months
  Will be treated as a continuous variable and will be summarized by treatment group and time-point using the mean, median, standard deviation, and the appropriate percentiles. The effectiveness of the RMT program on each respiratory outcome will be assessed by comparing the preoperative change between groups using an ANCOVA model, with an adjustment for the pretreatment levels. For each outcome, the preoperative change (T1-T0) will be modeled as a function of treatment group (RMT versus usual care) and pre-treatment levels. A one-sided Wald type-test about coefficient for treatment group will evaluate whether the RMT program had a beneficial impact on the given respiratory outcome. All model assumptions will be verified graphically using quantile-quantile and residual plots. Transformations will be applied as appropriate.
Change in peak exercise capacity (VO2peak) | Baseline up to 12 months
  Will be treated as a continuous variable and will be summarized by treatment group and time-point using the mean, median, standard deviation, and the appropriate percentiles. The effectiveness of the RMT program on each respiratory outcome will be assessed by comparing the preoperative change between groups using an ANCOVA model, with an adjustment for the pretreatment levels. For each outcome, the preoperative change (T1-T0) will be modeled as a function of treatment group (RMT versus usual care) and pre-treatment levels. A one-sided Wald type-test about coefficient for treatment group will evaluate whether the RMT program had a beneficial impact on the given respiratory outcome. All model assumptions will be verified graphically using quantile-quantile and residual plots. Transformations will be applied as appropriate.

SECONDARY OUTCOMES:
Metabolic and muscle physiology marker analysis | At time of surgical resection
  Assays of muscle biopsies will be performed for metabolic and muscle physiology markers. The correlative markers will be compared between RMT responders, RMT non-responders, and usual care (control) in a pairwise fashion using Holm-Bonferroni adjusted t-tests. Responders will be those who present with a > 15% increase in inspiratory and expiratory muscle strength. The gene-level raw count values of micro ribonucleic acid (mRNA)s will be analyzed with the edgeR Bioconductor package in R, first for normalization with the trimmed mean of M-values method, and then for comparison of expression between treatments using generalized linear models with negative binomial distribution and a likelihood ratio test to generate p values. False discovery rates (FDR) will be estimated from p-values with the Benjamini-Hochberg method, and mRNAs/genes with FDR < 0.05 and fold-change values of >= 1 log2 unit will be considered as differentially expressed.
Gene expression ribonucleic acid (RNA) extraction, reverse transcription, and real-time quantitative polymerase chain reaction (PCR) analysis | At time of surgical resection
  Assays of muscle biopsies will be performed for gene expression of RNA extraction, reverse transcription and real-time PCR. The correlative markers will be compared between RMT responders, RMT non-responders, and usual care (control) in a pairwise fashion using Holm-Bonferroni adjusted t-tests. Responders will be those who present with a > 15% increase in inspiratory and expiratory muscle strength. The gene-level raw count values of mRNAs will be analyzed with the edgeR Bioconductor package in R, first for normalization with the trimmed mean of M-values method, and then for comparison of expression between treatments using generalized linear models with negative binomial distribution and a likelihood ratio test to generate p values. FDR will be estimated from p-values with the Benjamini-Hochberg method, and mRNAs/genes with FDR < 0.05 and fold-change values of >= 1 log2 unit will be considered as differentially expressed.
Change in quality of life (QoL) | Baseline up to 12 months
  Will be measured by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) - Core (C)30. The QoL measures are treated as continuous and will be summarized by treatment group and time-point using the mean, median, standard deviation, and the appropriate percentiles. The change in QoL measures (from baseline) will be modeled as a function of treatment group, time-point, their two-way interaction, and baseline levels using a general linear model. Comparisons of QoL at each time-point will utilize Holm-Bonferroni adjusted tests about the appropriate contrasts of model estimates. All model assumptions will be verified graphically using quantile-quantile and residual plots. Transformations will be applied as appropriate.
Change in QoL | Baseline up to 12 months
  Will be measured by EORTC QLQ - Lung Cancer 13. The QoL measures are treated as continuous and will be summarized by treatment group and time-point using the mean, median, standard deviation, and the appropriate percentiles. The change in QoL measures (from baseline) will be modeled as a function of treatment group, time-point, their two-way interaction, and baseline levels using a general linear model. Comparisons of QoL at each time-point will utilize Holm-Bonferroni adjusted tests about the appropriate contrasts of model estimates. All model assumptions will be verified graphically using quantile-quantile and residual plots. Transformations will be applied as appropriate.
Change in fatigue level | Baseline up to 12 months
  Will be measured by Functional Assessment of Chronic Illness Therapy Fatigue. The QoL measures are treated as continuous and will be summarized by treatment group and time-point using the mean, median, standard deviation, and the appropriate percentiles. The change in QoL measures (from baseline) will be modeled as a function of treatment group, time-point, their two-way interaction, and baseline levels using a general linear model. Comparisons of QoL at each time-point will utilize Holm-Bonferroni adjusted tests about the appropriate contrasts of model estimates. All model assumptions will be verified graphically using quantile-quantile and residual plots. Transformations will be applied as appropriate.
Change in sleepiness (sleep apnea) | Baseline up to 12 months
  Will be measured by the Epworth Sleepiness Scale. The QoL measures are treated as continuous and will be summarized by treatment group and time-point using the mean, median, standard deviation, and the appropriate percentiles. The change in QoL measures (from baseline) will be modeled as a function of treatment group, time-point, their two-way interaction, and baseline levels using a general linear model. Comparisons of QoL at each time-point will utilize Holm-Bonferroni adjusted tests about the appropriate contrasts of model estimates. All model assumptions will be verified graphically using quantile-quantile and residual plots. Transformations will be applied as appropriate.
Change in sleepiness (sleep apnea) | Baseline up to 12 months
  Will be measured by the Stop-Bang Questionnaire. The QoL measures are treated as continuous and will be summarized by treatment group and time-point using the mean, median, standard deviation, and the appropriate percentiles. The change in QoL measures (from baseline) will be modeled as a function of treatment group, time-point, their two-way interaction, and baseline levels using a general linear model. Comparisons of QoL at each time-point will utilize Holm-Bonferroni adjusted tests about the appropriate contrasts of model estimates. All model assumptions will be verified graphically using quantile-quantile and residual plots. Transformations will be applied as appropriate.
Change in sleep quality | Baseline up to 12 months
  Will be measured by Pittsburgh Sleep Quality Index. The QoL measures are treated as continuous and will be summarized by treatment group and time-point using the mean, median, standard deviation, and the appropriate percentiles. The change in QoL measures (from baseline) will be modeled as a function of treatment group, time-point, their two-way interaction, and baseline levels using a general linear model. Comparisons of QoL at each time-point will utilize Holm-Bonferroni adjusted tests about the appropriate contrasts of model estimates. All model assumptions will be verified graphically using quantile-quantile and residual plots. Transformations will be applied as appropriate.
Change in anxiety and depression | Baseline up to 12 months
  Will be measured by Hospital Anxiety and Depression Scale. The QoL measures are treated as continuous and will be summarized by treatment group and time-point using the mean, median, standard deviation, and the appropriate percentiles. The change in QoL measures (from baseline) will be modeled as a function of treatment group, time-point, their two-way interaction, and baseline levels using a general linear model. Comparisons of QoL at each time-point will utilize Holm-Bonferroni adjusted tests about the appropriate contrasts of model estimates. All model assumptions will be verified graphically using quantile-quantile and residual plots. Transformations will be applied as appropriate.
Change in dyspnea | Baseline up to 12 months
  Will be measured by the Borg Dyspnea Scale. The QoL measures are treated as continuous and will be summarized by treatment group and time-point using the mean, median, standard deviation, and the appropriate percentiles. The change in QoL measures (from baseline) will be modeled as a function of treatment group, time-point, their two-way interaction, and baseline levels using a general linear model. Comparisons of QoL at each time-point will utilize Holm-Bonferroni adjusted tests about the appropriate contrasts of model estimates. All model assumptions will be verified graphically using quantile-quantile and residual plots. Transformations will be applied as appropriate.
Presence or absence of pneumonia diagnoses | Up to 12 months
  Pneumonia status is treated as dichotomous data and will be summarized by treatment group using frequencies and relative frequencies. The pneumonia rates will be compared between treatment groups using a one-sided Fisher exact test, as we expect the RMT program to reduce rates.

OTHER OUTCOMES:
Total hospital length of stay (LOS) | Up to 12 months
  Will be treated as continuous data and will be summarized by treatment group using the mean, median, standard deviation, and the appropriate percentiles. Comparisons between treatment groups will be made using one-sided t-tests or Mann-Whitney U tests (as appropriate).
Total intensive care unit LOS | Up to 12 months
  Will be treated as continuous data and will be summarized by treatment group using the mean, median, standard deviation, and the appropriate percentiles. Comparisons between treatment groups will be made using one-sided t-tests or Mann-Whitney U tests (as appropriate).
Pre-operative LOS | From date of admission to the date of surgery
  Will be treated as continuous data and will be summarized by treatment group using the mean, median, standard deviation, and the appropriate percentiles. Comparisons between treatment groups will be made using one-sided t-tests or Mann-Whitney U tests (as appropriate).
Lung infection rates | Up to 12 months
  Lung infection will be treated as dichotomous data and will be summarized by treatment group using frequencies and relative frequencies. Comparison of infection rates between treatment groups will be made using Fisher?s exact test.
Identified molecular marker analysis | Up to 1 month post-surgery
  Analysis of identified molecular markers will be completed to correlate with patient outcome and potentially differentiate responders from non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Saikrishna S Yendamuri, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States